CLINICAL TRIAL: NCT04017741
Title: A Phase IV Single Blind Placebo-controlled Cross Over Study to Investigate the Efficacy of Greater Occipital Nerve Block With Local Anesthetic and Steroid in Patients With Chronic Migraine
Brief Title: A Study Investigating the Efficacy of GON Blocks.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 009665 BLT
Record Dates: First submitted 2019-04-16; First posted 2019-07-12 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2019-11

CONDITIONS: Migraine; Chronic Migraine, Headache
Keywords: Chronic migraine, GON blocks
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Lidocaine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: Consented participants will be individually randomised by the Principal Investigator (PI) in a 1:1 ratio to receive either the GON block (active group) or the placebo injection (control group).
Who Masked: Participant, Investigator
Masking Description: This is a blinded, placebo controlled study, whereby the patient and the research team except for the injector are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active group (Active Comparator): The active group will be administered 2 mls of 2% lidocaine and 80mg methylprednisolone.
  Interventions: Drug: Combined Depo-Medrone and Lidocaine; Drug: Sodium Chloride 0.9% Inj
- Placebo group (Placebo Comparator): The placebo group will be administered 4mls of 0.9% saline.
  Interventions: Drug: Combined Depo-Medrone and Lidocaine; Drug: Sodium Chloride 0.9% Inj

INTERVENTIONS:
Drug: Combined Depo-Medrone and Lidocaine — Patients will be randomised 1:1 to receive the active or placebo arm. The nerve is located along the superior nuchal line, where it bilaterally lies medial to the occipital artery. The scalp is prepped with alcohol and using 23G needle, the IMPs are injected at a 90 degrees angle till the bony endpoint is obtained. A combination of 2 mls of 2% lidocaine and 80mg methylprednisolone will be administered.
  Patients who no longer receive any benefit will be crossed over to the placebo arm.
  Other Names: Methylprednisolone Acetate BP 40mg/mL:; Lidocaine Hydrochloride 2%:
Drug: Sodium Chloride 0.9% Inj — Patients will be randomised 1:1 to receive the active or placebo arm. The nerve is located along the superior nuchal line, where it bilaterally lies medial to the occipital artery. The scalp is prepped with alcohol and using 23G needle the 4mls of normal saline (0.9%) are injected at a 90 degrees angle till the bony endpoint is obtained. Patients who no longer receive any benefit will be crossed over to the active arm.
  Other Names: normal saline 0.9%

SUMMARY:
Greater occipital nerve block ("GON block") is carried out extensively in the treatment of chronic migraine, but more research is required to understand the effectiveness of the procedure. It consists of a superficial injection of local anaesthetic and steroid around a nerve at the back of the head that supplies sensation to part of the scalp. This study intends to provide more detailed information on the effectiveness, safety and tolerability of GON block with local anaesthetic and steroid in patients with chronic migraine. It does this by comparing it to a dummy (placebo) procedure (a needle is inserted near the nerve, but no therapeutic substance is injected). It is a "cross-over study": all patients will receive both the GON block and the dummy procedure (not necessarily in that order), with a period in between to assess the response to the first injection. The GON block will entail an injection of 2 mls of 2% lidocaine (a local anaesthetic) and 80 mg of DepoMedrone (a steroid) through a fine needle (a total of 4 mls). The dummy procedure will consist of an injection of 4 mls of normal saline (a solution of common salt and water) through a fine needle. Patients will be followed up at various time points throughout 6 months whilst being enrolled on the study.

DETAILED DESCRIPTION:
Chronic migraine is characterised by frequency of headache ≥ 15 days per month for more than 3 months. The location can be unilateral or bilateral. Usually described as pulsating in nature, it may be aggravated by, or cause avoidance of, routine activities of daily living. There can be associated light and noise sensitivity. Greater occipital nerve (GON) blockade with local anaesthetics and steroids has been used as a preventative strategy for a range of headaches including, migraine, cluster headache and hemicrania continua.

The occipital nerves have a sensory distribution in the occipital area. The greater occipital nerve derives most of its fibres from the C2 dorsal root [6]. It passes over the superior nuchal line, mid-way between the mastoid process and the occipital protuberance, just lateral to the insertion of the nuchal ligaments. The lesser occipital nerve passes lateral to the greater occipital nerve, over the nuchal ridge. Although the exact mechanism of action remains unclear, injection of steroid in the vicinity of GON nerve can have both a local effect (decreasing nociception) and a delayed central nociceptive response, possibly through an action on trigeminocervical relay

Although GON block is carried out extensively in the prophylaxis of chronic migraine, the evidence remains equivocal. In the UK, the National Institute for Clinical Excellence have yet to include GON blocks in their guidance and protocols on the treatment of both chronic headache and migraine. This randomised, single-blinded, placebo-controlled multicentre cross-over study intends to assess the efficacy, safety and tolerability of greater occipital nerve block with local anaesthetic and steroid in patients with chronic migraine with the primary objective to investigate any improvement in disability associated with chronic migraine disorder. We also intend to identify any economic outcomes associated with these injections in the management of chronic migraine.

GON block with local anaesthetic and steroid for chronic migraine and the placebo procedure will be performed in the outpatient setting. They will be carried out only by appropriately qualified members of the research team adhering to strict aseptic conditions and following standard operating protocols with regards to admission and discharge criteria in the outpatient settings.

GON block is routinely carried out in the UK and poses minimal risks to the patient. Although GON block is carried out extensively in prophylaxis of chronic migraine, the evidence remains equivocal. In the UK, the National Institute for Health and Care Excellence (NICE) have yet to include GON blocks in their guidance and protocols on the treatment of both chronic headache and migraine.

The aim of this study is to assess the efficacy, safety and tolerability of greater occipital nerve block with local anaesthetic and steroid in patients with chronic migraine of more than three months' duration.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over the age of 18 who are able to provide a written consent
* Ability to read and write English, due to questionnaire use in study
* Diagnosis of chronic migraine with or without acute relief medication overuse (ICHD-III codes 1.3 and 8.2); as confirmed by diary documentation (headache on 15 or more days a month for at least 3 months)

Exclusion Criteria:

* Patient refusal
* Participation in any trial of any investigational products or interventional research project within the previous eight weeks to enrolment
* Patients unable to commit to the six-month study duration (PI judgment)
* Any known contraindication(s) to the IMPs as described by the manufacturer's Summary of Product Characteristics (SmPCs)
* Patients with a history of substance abuse
* Pregnant or breastfeeding patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
The changes in disability associated with chronic migraine disorder at baseline | Baseline
  The average change in HIT-6 scores which measures six patient self-assessment-questions and helps distinguish the impact the effect of headache and its treatment on the patient's functional status and quality of life.
The changes in baseline headache impact test scores (HIT-6) at 4 weeks | 4 weeks
  The average change in HIT-6 scores which measures six patient self-assessment-questions and helps distinguish the impact the effect of headache and its treatment on the patient's functional status and quality of life.
The changes in baseline headache impact test scores (HIT-6) at 8 weeks | 8 weeks
  The average change in HIT-6 scores which measures six patient self-assessment-questions and helps distinguish the impact the effect of headache and its treatment on the patient's functional status and quality of life.
The changes in baseline headache impact test scores (HIT-6) at 12 weeks | 12 weeks
  The average change in HIT-6 scores which measures six patient self-assessment-questions and helps distinguish the impact the effect of headache and its treatment on the patient's functional status and quality of life.
The changes in baseline headache impact test scores (HIT-6) at 16 weeks | 16 weeks
  The average change in HIT-6 scores which measures six patient self-assessment-questions and helps distinguish the impact the effect of headache and its treatment on the patient's functional status and quality of life.
The changes in baseline headache impact test scores (HIT-6) at 20 weeks | 20 weeks
  The average change in HIT-6 scores which measures six patient self-assessment-questions and helps distinguish the impact the effect of headache and its treatment on the patient's functional status and quality of life.
The changes in baseline headache impact test scores (HIT-6) at 24 weeks | 24 weeks
  The average change in HIT-6 scores which measures six patient self-assessment-questions and helps distinguish the impact the effect of headache and its treatment on the patient's functional status and quality of life.
change in quality of life relating to migraine at baseline | baseline
  average change MSQ (Migraine Specific Quality of Life Questionnaire) to assess quality of life relating to migraine. MSQ Version 2.1 consists of 14 questions.
change in quality of life relating to migraine from baseline at 4 weeks | 4 weeks
  average change MSQ (Migraine Specific Quality of Life Questionnaire) to assess quality of life relating to migraine. MSQ Version 2.1 consists of 14 questions.
change in quality of life relating to migraine from baseline at 8 weeks | 8 weeks
  average change MSQ (Migraine Specific Quality of Life Questionnaire) to assess quality of life relating to migraine. MSQ Version 2.1 consists of 14 questions.
change in quality of life relating to migraine from baseline at 12 weeks | 12 weeks
  average change MSQ (Migraine Specific Quality of Life Questionnaire) to assess quality of life relating to migraine. MSQ Version 2.1 consists of 14 questions.
change in quality of life relating to migraine from baseline at 16 weeks | 16 weeks
  average change MSQ (Migraine Specific Quality of Life Questionnaire) to assess quality of life relating to migraine. MSQ Version 2.1 consists of 14 questions.
change in quality of life relating to migraine from baseline at 20 weeks | 20 weeks
  average change MSQ (Migraine Specific Quality of Life Questionnaire) to assess quality of life relating to migraine. MSQ Version 2.1 consists of 14 questions.
change in quality of life relating to migraine from baseline at 24 weeks | 24 weeks
  average change MSQ (Migraine Specific Quality of Life Questionnaire) to assess quality of life relating to migraine. MSQ Version 2.1 consists of 14 questions.
change in health related quality of life associated with chronic migraine disorder at baseline | baseline
  The changes reported in the short form survey with 12 questions (SF-12), comprised of two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life.
change in health related quality of life associated with chronic migraine disorder from baseline at 4 weeks | 4 weeks
  The changes reported in the short form survey with 12 questions (SF-12), comprised of two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life.
change in health related quality of life associated with chronic migraine disorder from baseline at 8 weeks | 8 weeks
  The changes reported in the short form survey with 12 questions (SF-12), comprised of two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life.
change in health related quality of life associated with chronic migraine disorder from baseline at 12 weeks | 12 weeks
  The changes reported in the short form survey with 12 questions (SF-12), comprised of two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life.
change in health related quality of life associated with chronic migraine disorder from baseline at 16 weeks | 16 weeks
  The changes reported in the short form survey with 12 questions (SF-12), comprised of two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life.
change in health related quality of life associated with chronic migraine disorder from baseline at 20 weeks | 20 weeks
  The changes reported in the short form survey with 12 questions (SF-12), comprised of two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life.
change in health related quality of life associated with chronic migraine disorder from baseline at 24 weeks | 24 weeks
  The changes reported in the short form survey with 12 questions (SF-12), comprised of two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life.

SECONDARY OUTCOMES:
Change in Headache frequency & Severity at baseline | baseline
  changes in Frequency and severity as scored in the HIT-6 questionnaire. Total scores can range between 36-78. Scores higher than 60 can indicate more greater impact on patient life.
Change from baseline Headache frequency & Severity at 4 weeks | 4 weeks
  changes in Frequency and severity as scored in the HIT-6 questionnaire when compared to baseline. Total scores can range between 36-78. Scores higher than 60 can indicate more greater impact on patient life.
Change from baseline Headache frequency & Severity at 8 weeks | 8 weeks
  changes in Frequency and severity as scored in the HIT-6 questionnaire when compared to baseline. Total scores can range between 36-78. Scores higher than 60 can indicate more greater impact on patient life.
Change from baseline Headache frequency & Severity at 12 weeks | 12 weeks
  changes in Frequency and severity as scored in the HIT-6 questionnaire when compared to baseline. Total scores can range between 36-78. Scores higher than 60 can indicate more greater impact on patient life.
Change from baseline Headache frequency & Severity at 16 weeks | 16 weeks
  changes in Frequency and severity as scored in the HIT-6 questionnaire. Total scores can range between 36-78. Scores higher than 60 can indicate more greater impact on patient life.
Change in Headache frequency & Severity at 20 weeks | 20 weeks
  changes in Frequency and severity as scored in the HIT-6 questionnaire when compared to baseline.Total scores can range between 36-78. Scores higher than 60 can indicate more greater impact on patient life.
Change from baseline Headache frequency & Severity at 24 weeks | 24 weeks
  changes in Frequency and severity as scored in the HIT-6 questionnaire. Total scores can range between 36-78. Scores higher than 60 can indicate more greater impact on patient life.
Change in anxiety and depression levels at baseline | baseline
  Change in Hospital Anxiety and Depression Scores (HADS) questionnaire Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The higher the score, the more impact the headache has on the patient's life.
Change from baseline anxiety and depression levels at 4 weeks | 4 weeks
  Change in Hospital Anxiety and Depression Scores (HADS) questionnaire when compared to baseline. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The higher the score, the more impact the headache has on the patient's life.
Change from baseline anxiety and depression levels at 8 weeks | 8 weeks
  Change in Hospital Anxiety and Depression Scores (HADS) questionnaire when compared to baseline
Change from baseline anxiety and depression levels at 12 weeks | 12 weeks
  Change in Hospital Anxiety and Depression Scores (HADS) questionnaire when compared to baseline. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The higher the score, the more impact the headache has on the patient's life.
Change from baseline anxiety and depression levels at 16 weeks | 16 weeks
  Change in Hospital Anxiety and Depression Scores (HADS) questionnaire when compared to baseline. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The higher the score, the more impact the headache has on the patient's life.
Change from baseline anxiety and depression levels at 20 weeks | 20 weeks
  Change in Hospital Anxiety and Depression Scores (HADS) questionnaire when compared to baseline. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The higher the score, the more impact the headache has on the patient's life.
Change from baseline anxiety and depression levels at 24 weeks | 24 weeks
  Change in Hospital Anxiety and Depression Scores (HADS) questionnaire when compared to baseline. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The higher the score, the more impact the headache has on the patient's life.

CONTACTS AND LOCATIONS:
Overall Officials: Anish Bahra, Principal Investigator — University College London Hospital
Locations (1):
- Barts Health NHS Trust, London, United Kingdom